CLINICAL TRIAL: NCT02674516
Title: The Effect of Repeated Transcranial Direct Current Stimulation of the Prefrontal Cortex on Antisocial and Aggressive Behavior
Brief Title: The Effect of Repeated Prefrontal Cortex Stimulation on Antisocial and Aggressive Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 823967
Record Dates: First submitted 2016-01-26; First posted 2016-02-04 (Estimated); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Antisocial Behavior; Aggression
Keywords: antisocial behavior; aggression; transcranial direct current stimulation; dorsolateral prefrontal cortex; associated risk factors
MeSH Terms: conditions — Antisocial Personality Disorder; Aggression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anodal stimulation (Experimental): Participants in the active stimulation group will undergo 3 sessions of anodal bilateral transcranial direct stimulation (tDCS) of the dorsolateral prefrontal cortex (DLPFC) on three consecutive days. tDCS will be delivered by a battery-driven, constant-current stimulator connected to three saline-soaked surface sponge electrodes. Two anodal electrodes (25cm2) will be placed over the DLPFC bilaterally and one cathodal electrode (35cm2) will be placed at the back of the neck. Scalp electrodes will be positioned over the F3 and F4 according to the 10-20 EEG international system. A current of 2mA (1mA at each DLPFC site) will be applied for 20 minutes and the current will be ramped up and down at the beginning and end of the stimulation period.
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): The sham transcranial direct current stimulation condition will involve the same placement of the electrodes, current intensity, and ramp time as the real tDCS condition, but stimulation will only last for 30 seconds.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation
  Arms: Anodal stimulation
Device: Sham transcranial direct current stimulation
  Arms: Sham stimulation

SUMMARY:
This study investigates the relationship between prefrontal cortex activity and antisocial and aggressive behavior, and risk factors for such behavior. In the double-blind, randomized controlled trial, participants will undergo three sessions of anodal transcranial direct current stimulation of the dorsolateral prefrontal cortex or sham stimulation and complete survey and laboratory measures assessing antisocial behavior and risk factors. Heart rate and skin conductance will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Able to understand the nature of the study and give informed consent

Exclusion Criteria:

* Currently consuming anti-convulsant, anti-psychotic, or sedative/hypnotic medications
* Currently consuming anti-depressants
* History of seizures
* Metallic implants on the scalp
* Participation in other transcranial magnetic stimulation (TMS) or tDCS experiments on the same day
* History of adverse reactions to tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Raine, DPhil, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Anodal Stimulation: Participants in the active stimulation group will undergo 3 sessions of anodal bilateral transcranial direct stimulation (tDCS) of the dorsolateral prefrontal cortex (DLPFC) on three consecutive days. tDCS will be delivered by a battery-driven, constant-current stimulator connected to three saline-soaked surface sponge electrodes. Two anodal electrodes (25cm2) will be placed over the DLPFC bilaterally and one cathodal electrode (35cm2) will be placed at the back of the neck. Scalp electrodes will be positioned over the F3 and F4 according to the 10-20 EEG international system. A current of 2mA (1mA at each DLPFC site) will be applied for 20 minutes and the current will be ramped up and down at the beginning and end of the stimulation period.
  Transcranial direct current stimulation
- Sham Stimulation: The sham transcranial direct current stimulation condition will involve the same placement of the electrodes, current intensity, and ramp time as the real tDCS condition, but stimulation will only last for 30 seconds.
  Sham transcranial direct current stimulation
Period: Overall Study
Arm/Group | Anodal Stimulation | Sham Stimulation
Started | 17 | 15
Completed | 13 | 11
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Protocol Violation | 0 | 4
Not completed — Knowledge of study hypothesis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anodal Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.15 (10.77) | 33.27 (14.10) | 32.13 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 6 | 4 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Pins Inserted Into a Virtual Voodoo Doll After 48 Hours
Description: The number of pins (between 0 and 51) that participants decide to insert into a picture of a voodoo doll on a computer that represents either a romantic partner or close friend will be recorded.
Time Frame: On average, 48 hours after the first 20-minute tDCS or sham session ends
Measure: Mean (Standard Deviation); unit: pins
Arm/Group | Anodal Stimulation | Sham Stimulation
Number analyzed (Participants) | 13 | 11
pins | 3.77 (8.88) | .64 (1.50)

ADVERSE EVENTS:
Time Frame: 48 hours after the end of the first stimulation session
Arm/Group | Anodal Stimulation | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 12/13 | 8/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anodal Stimulation (N=13) | Sham Stimulation (N=11)
Itchiness (Skin and subcutaneous tissue disorders) | 12 (12) | 4 (4)
Lightheadedness (General disorders) | 3 (3) | 1 (1)
Pain (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Burning (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (4)
Mild warmth (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Pinching (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Iron taste (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT02674516/Prot_SAP_000.pdf